CLINICAL TRIAL: NCT00836602
Title: Placebo-Controlled, Ascending, Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-779788 in Healthy Subjects
Brief Title: Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-779788 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CV197-002
Record Dates: First submitted 2009-01-30; First posted 2009-02-04 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2009-08

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — 2-(2-(1-(2-chlorophenyl)-1-methylethyl)-1-(3'-(methylsulfonyl)-4-biphenylyl)-1H-imidazol-4-yl)-2-propanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- BMS-779788 or Placebo (Arm 1) (Active Comparator)
  Interventions: Drug: BMS-779788; Drug: Placebo
- BMS-779788 or Placebo (Arm 2) (Active Comparator)
  Interventions: Drug: BMS-779788; Drug: Placebo
- BMS-779788 or Placebo (Arm 3) (Active Comparator)
  Interventions: Drug: BMS-779788; Drug: Placebo

INTERVENTIONS:
Drug: BMS-779788 — Oral Solution, Oral, 1 mg, Once daily, 7 days
  Arms: BMS-779788 or Placebo (Arm 1)
Drug: BMS-779788 — Oral Solution, Oral, 2 mg, Once daily, 7 days
  Arms: BMS-779788 or Placebo (Arm 2)
Drug: BMS-779788 — Oral Solution, Oral, <= 4 mg, Once daily, 7 days
  Arms: BMS-779788 or Placebo (Arm 3)
Drug: Placebo — Oral Solution, Oral, 0 mg, Once daily, 7 days

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of multiple oral doses of BMS-779788 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Men and women (not of child bearing potential) ages 18 to 45
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Exclusion Criteria:

* Women of child bearing potential
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety assessment, including medical review of adverse event reports and the results of vital sign measurements, ECGs, physical examinations, and clinical laboratory tests | 8 times within 27 days of the first dose

SECONDARY OUTCOMES:
Pharmacokinetics (Target gene expression of BMS-779788 in whole blood and adipose tissue and corresponding serum markers) | After each dose panel

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Heidelberg, Victoria, Australia

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx